CLINICAL TRIAL: NCT03515447
Title: Romiplostim as a Platelet-transfusion Saving Strategy After Thoracic Transplantation and Circulatory or Respiratory Assistance Devices: A Before-after Study of 172 Patients
Brief Title: Romiplostim in Thoracic Transplantation
Acronym: N-PLATE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0044
Record Dates: First submitted 2018-03-21; First posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Thrombocytopenia
Keywords: transfusion saving strategy; heart or lung transplantation; assist device; Extra Corporal Life Support (ECLS); Left Ventricular Assist Device (LVAD ); Total artificial Heart
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before period: During this period no patient received Romiplostim.
- After period: Application of the transfusion saving strategy protocol through Romiplostim treatment.
  The first subcutaneous injection of 1.5 to 2 µg/kg of romiplostim was administered in the post-operative periods. An algorithm based on patient weight and platelet count was established to determine romiplostim doses. One injection per week was performed. Romiplostim posology was adjusted between 2 and 5µg/kg every week according to platelet count with a maximum of 4 administrations in the ICU.
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study
  Groups: After period

SUMMARY:
The investigators developed a platelet transfusion saving strategy based on thrombopoietin administration in heart or lung transplantation (HLT) patients or assist device implantation in bridge-to-transplantation (BTT) or bridge to-decision (BTD). This strategy was applied from May 2014 to October 2015 in patients whose platelet counts were below 100 Giga per liter (G/L). As part of a health care quality improvement project, the investigators evaluated this strategy in a before/after design. January 2010 to December 2013 constituted the before period.

DETAILED DESCRIPTION:
In may 2014, after Heart or Lung transplantation or assist device implantation, the investigators decided to off-label administered Romiplostim in patients with thrombocytopenia below 100 Giga per liter. The purpose was to reduce platelets transfusion side effects. Romiplostim was used off treatment algorithm was based on previously published data in idiopathic, thrombocytopenia, cirrhotic and hematological patients. The first subcutaneous injection of 1.5 to 2 μg/kg of romiplostim was administered in the postoperative periods. An algorithm based on patient weight and platelet count evolution was established to determine romiplostim doses to administered weekly. Romiplostim posology was adjusted between 2 and 5μg/kg according to platelet count with a maximum of 4 administrations in the ICU. If platelets remained below 50 Giga per liter after 2 injections, bone marrow analysis after hematologist referral was discussed. Platelet count until day 15 after the last injection was monitored to detect thrombocytosis.

In January 2016, the investigators decided to retrospectively assess Romiplostim implementation in the standard of care in the ICU through a Healthcare quality improvement project in a before/after design.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in ICU after HLT, BTT or BTD assist device implantation with platelet counts below 100G/L at least once in the post-operative period

Exclusion Criteria:

* age under 18 or over 65, combined heart and lung transplantation, multiple organ dysfunction syndrome (MODS), pericardial effusion, active surgical bleeding, assist device dysfunction or suspected/diagnosed heparin-induced thrombocytopenia. We also excluded patients with myelodysplastic or myeloproliferative syndrome, hematological malignancy, severe liver cirrhosis with a Child-Pugh score superior to 6, receiving antiplatelet therapy, aplasia diagnosed on bone marrow analyses, pregnancy, thrombophilia, prior pulmonary embolism or stroke in the previous 6 months. Thrombophilia was defined as factor V Leyden mutation, activated protein C resistance, protein S deficiency, protein C deficiency, prothrombin gene mutation, factor VIII excess, ATIII deficiency or antiphospholipid syndrome. For the assistance population, the protocol also excluded destination-therapy devices or patients with transplantation contraindications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart or lung transplantation (HLT) patients or assist device implantation in bridge-to-transplantation or to-decision; with platelet counts below 100G/L at least once in the post-operative period
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Number of platelets concentrate | Until day 28
  Cumulative platelets concentrate from day 1 to day 28 after thoracic transplantation or assist device implantation.

SECONDARY OUTCOMES:
Number of unit of Fresh Frozen Plasma transfused until day 28. | Until day 28
  The data will be collected from the blood service data base.
Number of unit of Packed red blood cells transfused until day 28. | Until day 28
  The data will be collected from the blood service data base.
Number of unit of whole labile blood products until day 28. | Until day 28
  The data will be collected from the blood service data base.
Transfusion cost | Until 1 year
alloimmunisation (DSA or non-DSA) until 1 year | At day 15, day30, month3, month6 and one year
Worst grade of graft rejection until 1 year. | At day 15, day30, month3, month6 and one year
  Acute cellular rejection (ACR) and antibody mediated rejection (AMR) will be quoted. We will considered the worst rejection grade.
Thrombotic event in ICU (stroke, deep venous thrombosis and pulmonary embolism) | Thrombotic events will be assessed daily in ICU until ICU discharge, up to 28 days. Pulmonary embolism and stroke will be diagnosed by CT scan and deep venous thrombosis by Echo-doppler examination.
Length of stay in ICU | From ICU admission to ICU discharge, up to 90 days. If the patient dies in ICU, the length of stay in ICU will be calculated from ICU admission until death.
Mechanical ventilation duration | Will be assessed daily from admission to ICU discharge, up to 28 days.Mechanical ventilation stand for invasive ventilator support such as endotracheal intubation or tracheostomy.Each day began with invasive ventilator support will be recorded.
Mortality in ICU | At day 28 and day 90

CONTACTS AND LOCATIONS:
Overall Officials: Karim ASEHNOUNE, MD, PhD, Principal Investigator — Nantes University Hospital